CLINICAL TRIAL: NCT00646126
Title: Validation of the Use of Istope-Based Molecular Techniques for Malaria Control
Brief Title: Antimalarial Treatments for Clearing Low Density P. Falciparum and Its Impact on Malaria Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tropical Medicine Research Institute (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); International Atomic Energy Agency (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUD 6/025
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2005-08

CONDITIONS: Plasmodium Falciparum; Asymptomatic Parataemia; Sub Patent Parasitaemia
MeSH Terms: conditions — Malaria, Falciparum | interventions — Sulfadoxine; Pyrimethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 1:Active comparator sulfadoxine-pyrimethamine plus artesunate
  Interventions: Drug: Sulfadoxine / Pyrimethamine (SP) plus artesunate (AS)
- 2 (Placebo Comparator): 2:placebo comparator
  Interventions: Drug: placebo tablet similar to active drug in shape and size

INTERVENTIONS:
Drug: Sulfadoxine / Pyrimethamine (SP) plus artesunate (AS) — Standard three day regimen
  Arms: 1
Drug: placebo tablet similar to active drug in shape and size — Dosage similar to active drug(standard three days regimen)
  Arms: 2

SUMMARY:
The malaria parasite Plasmodium falciparum remains at sub-patent level throughout the dry season in areas of seasonal malaria transmission. Targeting this parasite reservoir before the transmission season could be a good strategy for malaria control. We are conducting a randomized double blind placebo controlled mass drug administration trial in eight village to clear the dry season low level parasitaemia with an ultimate aim of controlling malaria in eastern Sudan.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the 8 villages

Exclusion Criteria:

* Pregnancy
* History of allergy to sulfa drugs

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-08

PRIMARY OUTCOMES:
Parsitaemia detected during the transmission season among dry season PCR negative persons in the intervention and control villages | October to December 2006

SECONDARY OUTCOMES:
1. Malaria prevalence during the transmission season 2. Frequency of mutation in drug resistance genes

CONTACTS AND LOCATIONS:
Overall Officials: Badria B El Sayed, PhD,MSc,BSc, Principal Investigator — Tropical Medicine Research Institute
Locations (1):
- Tropical Medicine Research Institute, Khartoum, Khartoum State, Sudan

REFERENCES:
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740